CLINICAL TRIAL: NCT04690556
Title: A Global, Phase III, Double Blind, Randomized Controlled Study to Compare the Efficacy, Safety & Immunogenicity of LUBT010 With Lucentis® in Patients With Neovascular Age Related Macular Degeneration
Brief Title: Study to Compare Efficacy, Safety, and Immunogenicity of LUBT010 (Proposed Ranibizumab Biosimilar) and Lucentis® in Patients With Neovascular AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRP/LUBT010/2016/008; 2017-004409-42 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-12-30 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular age-related macular degeneration, Ranibizumab
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: LUBT010 (proposed ranibizumab biosimilar) (Experimental)
  Interventions: Drug: LUBT010 (proposed ranibizumab biosimilar)
- Drug: Lucentis (ranibizumab) (Active Comparator)
  Interventions: Drug: Lucentis (ranibizumab)

INTERVENTIONS:
Drug: LUBT010 (proposed ranibizumab biosimilar) — LUBT010 (proposed ranibizumab biosimilar) 0.5 mg via intravitreal injection once monthly
  Arms: Drug: LUBT010 (proposed ranibizumab biosimilar)
Drug: Lucentis (ranibizumab) — Lucentis® 0.5 mg via intravitreal injection once monthly
  Arms: Drug: Lucentis (ranibizumab)

SUMMARY:
This study is designed to compare the efficacy, safety and immunogenicity of LUBT010 with Lucentis® given as once monthly intravitreal injection in patients with neovascular age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This is a global, phase III, double blind, randomized controlled study to compare the efficacy, safety & immunogenicity of LUBT010 with Lucentis® in patients with neovascular age-related macular degeneration.

Eligible patients will be randomly assigned in 1:1 ratio to receive once monthly intravitreal injection of LUBT010 or Lucentis® for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory male or female participants with age ≥ 50 years at the time of screening
2. Capable of understanding and giving written informed consent
3. Primary or recurrent (anti-vascular endothelial growth factor naïve) active choroidal neovascularization (CNV) lesions involving the foveal center secondary to AMD
4. Best corrected visual acuity (BCVA) between 20/40 and 20/200 (Snellen equivalent) in the study eye, using ETDRS testing
5. Willingness and ability to undertake all scheduled visits and assessments

Exclusion Criteria:

1. Known hypersensitivity to ranibizumab or any of the components of study medication
2. Known history of allergy to fluorescein dye
3. Scar, fibrosis, or atrophy involving the center of the fovea in the study eye
4. Subretinal hemorrhage in the study eye that involves the center of the fovea
5. Uncontrolled glaucoma
6. Use of prohibited treatments

Other In-/Exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (6):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Bruce A. Segal, MD, PA, Delray Beach, Florida
  - Cumberland Valley Retina Consultants, P.C., Hagerstown, Maryland
  - UPMC Eye Center - Eye and Ear Institute, Pittsburgh, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Valley Retina Institute, McAllen, Texas
- Bulgaria (10):
  - Medical Center Oxycom EOOD, Burgas
  - Eye medical center - Visus, Gorna Oryahovitsa
  - University First MHAT-Sofia, St. Joan Krastitel EAD, Sofia
  - MC Ophta-Nevro, Sofia
  - Specialized Eye Hospital Pentagram, Sofia
  - DCC Alexandrovska, EOOD, Sofia
  - Military Medical Academy - MHAT, Sofia
  - Specialized Hospital for Active Treatment of Ophthalmologic Diseases Zora, OOD, Sofia
  - MHAT Trakia, EOOD, Stara Zagora
  - Medical Center Vereya EOOD, Stara Zagora
- Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr, Hungary
- India (40):
  - The Eye Care Center, Guwahati, Assam
  - Drishtipunj Eye Hospital Pvt Ltd, Patna, Bihar
  - Advance Retina Care, Ahmedabad, Gujarat
  - Sadguru Netra Chikitsalaya, Ahmedabad, Gujarat
  - Netralaya - Super Speciality Eye Hospital, Ahmedabad, Gujarat
  - Rising Retina Clinic, Ahmedabad, Gujarat
  - Government Eye Hospital M & J Institute of Ophthalmology, Ahmedabad, Gujarat
  - M & J Western Regional Institute of Ophthalmology, Ahmedabad, Gujarat
  - P N Desai Eye Hospital, Ahmedabad, Gujarat
  - Kanoria Hospital and Research Center, Gandhinagar, Gujarat
  - Shivam Retina Clinic and Eye Hospital, Surat, Gujarat
  - Kiran Hospital Multi Super Speciality Hospital & Research Centre, Surat, Gujarat
  - Kashyap Memorial Eye Hospital Pvt. Ltd., Ranchi, Jharkhand
  - Nethra Eye Hospital, Bangalore, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - JSS Hospital, Mysore, Karnataka
  - Regional Institute of Opthalmology, Trivandrum, Kerala
  - Deshmukh Eye Hospital, Amravati, Maharashtra
  - Kamalnayan Bajaj Hospital, Aurangabad, Maharashtra
  - Aditya Jyot Eye Hospital Pvt. Ltd., Mumbai, Maharashtra
  - Shroff Eye Hospital & Vision Research Centre, Mumbai, Maharashtra
  - Kenia Eye Hospital, Mumbai, Maharashtra
  - Anideep Eye Hospital, Mumbai, Maharashtra
  - Topiwala National Medical College & B. Y. L. Nair Charitable Hospital, Mumbai, Maharashtra
  - Ambade Eye Hospital, Nagpur, Maharashtra
  - Dhadiwal Hospital in Coalition with Shreeji Healthcare, Nashik, Maharashtra
  - Vijay Vallabh Hospital and Medical Research Center, Pālghar, Maharashtra
  - Dr. D. Y. Patil Medical College, Pune, Maharashtra
  - Insight Institute of Ophthalmology, Pune, Maharashtra
  - Sri Guru Ram Das Institute of Medical Sciences & Research, Amritsar, Punjab
  - Advanced Eye Centre Post Graduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Dr.Agarwal's Eye Hospital, Tirunelveli, Tamil Nadu
  - Dr. J L Rohatgi Memorial Eye Hospital, Kanpur, Uttar Pradesh
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Sam Eye Hospital, Lucknow, Uttar Pradesh
  - R.K.Netralaya Eye Hospital (P) Ltd., Varanasi, Uttar Pradesh
  - Regional Institute of Ophthalmology, Kolkata, West Bengal
  - Dr. Shroff's Charity Eye Hospital, New Delhi
  - Sir Ganga Ram Hosptial, New Delhi
  - Aakash Healthcare Super Specialty Hospital, New Delhi
- Poland (8):
  - Szpital Świętego Łukasza S. A., Bielsko-Biala
  - Specjalistyczny Osrodek Okulistyczny Oculomedica, Bydgoszcz
  - Prywatna Klinika Okulistyczna OFTALMIKA, Bydgoszcz
  - Provisus Badania Kliniczne Sp. z o.o., Częstochowa
  - Clinical Medical Research Sp. z o.o., Katowice
  - Gabinet Okulistyczny prof. Edward Wylegala, Katowice
  - ETG Lodz, Lodz
  - CaminoMed - Specjalistyczne Gabinety Lekarskie, Tarnowskie Góry
- Russia (5):
  - LLC HI Optic-Center, Chelyabinsk
  - RSHI State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - BHI of Omsk region Clinical Ophthalmology Hospital n.a V.P. Vykhodtsev, Omsk
  - Standard Clinic Penza LLC, Penza
  - LLC X7 Clinical research, Saint Petersburg
- Slovakia (8):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Nemocnica svateho Michala, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - Nemocnica Poprad a.s., Poprad
  - Nemocnica s poliklinikou Trebisov a.s., Trebišov
  - Fakultna nemocnica Trencin, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make Individual Participant Data (IPD) available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: [Not Specified]
Pre-assignment Details: [Not Specified]
Groups:
- LUBT010 (Proposed Ranibizumab Biosimilar); Lucentis (Ranibizumab): 0.5 mg via intravitreal injection once monthly
Period: Overall Study
Arm/Group | LUBT010 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Started | 299 | 301
Completed | 256 | 269
Not Completed | 43 | 32
Not completed — Adverse Event | 6 | 4
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 1 | 4
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 25 | 17
Not completed — Prohibited medications and other reasons | 3 | 1

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Total: Total of all reporting groups
Arm/Group | LUBT010 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab) | Total
Number analyzed (Participants) | 299 | 301 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8.75) | 73.5 (7.90) | 73.3 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 146 | 297
  Male | 148 | 155 | 303
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 158 | 147 | 305
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 141 | 153 | 294
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in BCVA From Baseline in the Study Eye at the End of 12 Months
Description: Early treatment diabetic retinopathy study (ETDRS) charts were used for visual acuity measurement
Time Frame: Baseline and 12 Months
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | LUBT010 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 295 | 296
Letters | 11.17 (0.689) | 11.14 (0.680)
Statistical Analysis 1: Comparison: LUBT010 (Proposed Ranibizumab Biosimilar) vs Lucentis (Ranibizumab); LUBT010 (Proposed Ranibizumab Biosimilar) - Lucentis; Test type: Equivalence — Therapeutic equivalence was assessed based on the two-sided 90% Confidence Interval (CI) of the difference in least squares mean changes in BCVA from baseline at month 12 between LUBT010 and Lucentis for the pre-defined equivalence margin of (-4 letters, 4 letters); Least squares mean difference = 0.03, 90% CI 2-sided [-1.52 to 1.58], Standard Error of Mean 0.945 — Therapeutic equivalence met

2. Secondary Outcome: Mean Change in BCVA From Baseline in the Study Eye at the End of 3 Months
Description: ETDRS charts were used for visual acuity measurement summarized descriptively by treatment arm and time point
Time Frame: Baseline and 3 Months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | LUBT010 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 295 | 296
Letters | 7.3 (8.38) | 6.6 (7.97)

3. Secondary Outcome: Mean Change in BCVA From Baseline in the Study Eye at the End of 6 Months
Description: ETDRS charts were used for visual acuity measurement summarized descriptively by treatment arm and time point
Time Frame: Baseline and 6 Months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | LUBT010 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 295 | 296
Letters | 9.5 (9.67) | 8.7 (10.35)

4. Secondary Outcome: Mean Change in BCVA From Baseline in the Study Eye at the End of 9 Months
Description: ETDRS charts were used for visual acuity measurement summarized descriptively by treatment arm and time point
Time Frame: Baseline and 9 Months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | LUBT010 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 295 | 296
Letters | 10.6 (11.36) | 10.4 (10.62)

ADVERSE EVENTS:
Time Frame: AE reporting extended from date of informed consent until Month 12 (EOS visit)
Description: All AEs (ocular or non-ocular) were recorded. A treatment-emergent AE (TEAE) was defined as an AE that began or worsened in severity after at least 1 dose of study drug was administered.
Arm/Group | LUBT010 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
All-Cause Mortality (participants affected / at risk) | 3/299 | 4/301
Serious Adverse Events (participants affected / at risk) | 26/299 | 23/301
Other Adverse Events (participants affected / at risk) | 21/299 | 26/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LUBT010 (Proposed Ranibizumab Biosimilar) (N=299) | Lucentis (Ranibizumab) (N=301)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0
Non-infectious endophthalmitis (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ulcerative gastritis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 0 | 1
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Tuberculin test positive (Investigations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LUBT010 (Proposed Ranibizumab Biosimilar) (N=299) | Lucentis (Ranibizumab) (N=301)
Neovascular age-related macular degeneration (Eye disorders) | 21 | 26

LIMITATIONS AND CAVEATS:
[Not Applicable]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT04690556/Prot_SAP_000.pdf